CLINICAL TRIAL: NCT01514331
Title: Determination of Ventilatory Parameters and Inflammatory Responses of Neonates Who Are Ventilated by Volume Guarantee Combined With Synchronized Intermittent Mandatory Ventilation or Pressure Support Ventilation
Brief Title: Ventilatory Parameters and Inflammatory Responses of Neonates Ventilated by Different Modes of Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Ebru Ergenekon, Prof.Dr, Gazi University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 01/2011-68
Record Dates: First submitted 2011-12-20; First posted 2012-01-23 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-11

CONDITIONS: Respiratory Distress, Newborn; Ventilator Induced Lung Injury
Keywords: Ventilator Induced Lung Injury; Neonatal respiratory distress; Mechanical ventilation
MeSH Terms: conditions — Pulmonary Atelectasis; Ventilator-Induced Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PSV+VG (Active Comparator): Neonates who require mechanical ventilation and randomised to pressure support + volume guarantee (PSV+VG) mode
  Interventions: Other: PSV+VG (pressure support ventilation+volume guarantee)
- SIMV+VG (Active Comparator): Neonates who require mechanical ventilation and randomised to synchronised intermittant mandatory ventilation + volume guarantee (SIMV+VG) mode
  Interventions: Other: SIMV+VG mode of ventilation (synchronized intermittent mandatory ventilation+volume guarantee)

INTERVENTIONS:
Other: SIMV+VG mode of ventilation (synchronized intermittent mandatory ventilation+volume guarantee) — Neonates who need mechanical ventilation will be ventilated with SIMV+VG mode
  Other Names: SIMV + VG mode of ventilation
  Arms: SIMV+VG
Other: PSV+VG (pressure support ventilation+volume guarantee) — Neonates who need mechanical ventilation will be ventilated with PSV+VG
  Other Names: PSV+ VG mode of ventilation
  Arms: PSV+VG

SUMMARY:
The main purpose of this study is to investigate effects of SIMV+VG (synchronized intermittent mandatory ventilation+volume guarantee) or PSV+VG (pressure support ventilation+volume guarantee) ventilation on vital signs, patient - mechanical ventilation synchrony, ventilation parameters and inflammatory mediators in neonates.

DETAILED DESCRIPTION:
Term or preterm neonates may need mechanical ventilation due to different etiologies. In all patients aim of mechanical ventilation is to promote pulmonary gas exchange, reduce the respiratory work of patient. Ideal mechanical ventilation must minimize pulmonary trauma with low inspiratory pressures that obtains adequate and constant tidal volumes. Ventilation associated pulmonary injury is an important subject that must be considered during mechanical ventilation. Atelectotrauma, volutrauma, barotrauma and biotrauma must be monitored. Volutrauma, barotrauma and oxygen toxicity cause cytokine increase that results in biotrauma. This parenchymal inflammation is a risk factor for chronic lung disease which is an important morbidity of ventilated neonates.

From past to present neonates were ventilated with different ventilation modes including IMV (Intermittent Mandatory Ventilation), SIMV, A/C (Assist Control Ventilation), PSV,HFV (High Frequency Ventilation). Both PSV and SIMV are patient trigger ventilation modes but SIMV is a time cycled and PSV is a flow cycled mode. In recent years hybrid techniques were developed to combine beneficial features of volume and pressure limited ventilation. In commercial ventilation devices these techniques have different names as volume guaranteed pressure limited ventilation (Drager Babylog 8000), pressure regulated volume controlled ventilation (Siemens servo 3000), volume guaranteed pressure support ventilation (VIP Bird Gold).

Since there is not a standard protocol for mechanical ventilation of neonates different countries and even different NICU's use different ventilation protocols.

Literature supports volume targetted ventilation to reduce barotrauma with low maximum inspiratory pressures and to reduce volutrauma with constant tidal volumes. When A/C+VG and SIMV+VG were compared in a crossover trial, more constant tidal volumes were obtained in A/C mode. Inflammatory cytokines have also been measured in different groups of patients with variable ventilatory management techniques. So far there has not been a randomized study published comparing VG+SIMV with VG+PSV in newborns with regards to tidal volume , peak inspiratory pressure variability,or inflammatory cytokines. Therefore in this study the investigators aimed to compare these two ventilation modes with regards to short term outcome.

ELIGIBILITY:
Inclusion Criteria:

* neonates with respiratory distress who need mechanical ventilation
* gestational age less than or equal to 37 weeks
* neonates who need mechanical ventilation within first 24 hours

Exclusion Criteria:

* neonates who need mechanical ventilation other than conventional ventilation

Max Age: 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2012-01; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
IL-1beta levels in tracheal aspirate material | Baseline and 72 hours of mechanical ventilation
  Tracheal aspirate will be analyzed for the mediator level and change from baseline will be reported
IL-6 level in tracheal aspirate | Baseline and 72 hours of mechanical ventilation
  Tracheal aspirate will be analyzed for IL6 level and the change from baseline will be reported
IL-8 in tracheal aspirate material | Baseline and 72 hours of mechanical ventilation
  Tracheal aspirate will be analyzed for the mediator level and change from baseline will be reported
IL-10 level in tracheal aspirate material | Baseline and 72 hours of mechanical ventilation
  Tracheal aspirate will be analyzed for the mediator level and change from baseline will be reported
TNF alfa in tracheal aspirate material | Baseline and 72 hours of mechanical ventilation
  Tracheal aspirate will be analyzed for the mediator level and change from baseline will be reported
tidal volume variability | 72 hours of mechanical ventilation or entire ventilation time if extubated earlier
  variability in tidal volume measured with babyview program
peak inspiratory pressure variability | 72 hours of mechanical ventilation or entire ventilation time if extubated earlier
  variability in peak inspiratory pressure measured with babyview program
respiratory rate variability | 72 hours of mechanical ventilation or entire ventilation time if extubated earlier
  changes in respiratory rate, tacypnea rate
oxygen saturation variability | 72 hours of mechanical ventilation or entire ventilation time if extubated earlier
  changes in oxygen saturation, desaturation rate, hyperoxy rate
lowest carbondioxide level (mmHg) | 72 hours of mechanical ventilation or entire ventilation time if extubated earlier
  ratio of hypocarbic blood gases and least pCo2 level
highest carbondioxide level (mmHg) | 72 hours of mechanical ventilation or entire ventilation time if extubated earlier
  ratio of hypercarbic blood gases and highest pCo2 level
lowest oxygen level (mmHg) | 72 hours of mechanical ventilation or entire ventilation time if extubated earlier
  ratio of hypoxic blood gases and least pO2 level
highest oxygen level (mmHg) | 72 hours of mechanical ventilation or entire ventilation time if extubated earlier
  ratio of hyperoxic blood gases and highest pO2 level

SECONDARY OUTCOMES:
bronchopulmonary dysplasia | 36 weeks corrected age
  Oxygen requirement at 36 weeks corrected age
patent ductus arteriosus | in the first week of post natal life of the patient
  Presence of hemodynamically significant patent ductus arteriosus in the first 7 days of life
necrotizing enterocolitis | 36 weeks corrected age
  Necrotising entercolitis defined by clinical and radiological findings
intraventricular hemorrhage | during first week
  Intraventricular hemorrhage diagnosed by head ultrasound
pneumothorax | during first 3 days
  Air leak diagnosed by chest x-ray
pulmonary interstitial emphysema | during first week
  Air leak diagnosed by x-ray
pulmonary hemorrhage | during first week
retinopathy of prematurity | until 36 weeks corrected age
  Retinal disease diagnosed by indirect opthtalmoscopic exam

CONTACTS AND LOCATIONS:
Overall Officials: Ebru N Ergenekon, MD, Principal Investigator — Gazi University, Division of newborn Medicine
Locations (1):
- Gazi University Hospital, Department of Pediatrics, Division of Newborn Medicine, Beşevler, Ankara, Turkey (Türkiye)